CLINICAL TRIAL: NCT00542347
Title: Comparison of the Gastric Acid Suppressive Effects of Esomeprazole and Generic Omeprazole
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Enrollment target not met due to high number of disqualified studies.
Sponsor: Queen's University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Adriana Lazarescu, GI Fellow, Queen's University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1054-07
Record Dates: First submitted 2007-10-09; First posted 2007-10-11 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Gastric Acid
Keywords: gastric acid; proton pump inhibitors; omeprazole; esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): * esomeprazole 20mg po once per day for 7 days
  * 24hr pH study on day 7
  * followed by washout for 7 days
  * generic omeprazole 20mg po once per day for 7 days
  * 24hr pH study on day 7
  Interventions: Drug: Esomeprazole first
- 2 (Active Comparator): * generic omeprazole 20mg po once per day for 7 days
  * 24hr pH study on day 7
  * followed by washout for 7 days
  * esomeprazole 20mg po once per day for 7 days
  * 24hr pH study on day 7
  Interventions: Drug: Generic omeprazole first

INTERVENTIONS:
Drug: Esomeprazole first — * esomeprazole 20mg po once per day for 7 days
  * 24hr pH study on day 7
  * followed by washout for 7 days
  * generic omeprazole 20mg po once per day for 7 days
  * 24hr pH study on day 7
  Arms: 1
Drug: Generic omeprazole first — * generic omeprazole 20mg po once per day for 7 days
  * 24hr pH study on day 7
  * followed by washout for 7 days
  * esomeprazole 20mg po once per day for 7 days
  * 24hr pH study on day 7
  Arms: 2

SUMMARY:
Proton pump inhibitors (PPI) are used to decrease stomach acid secretion. A generic form of omeprazole, one of the PPIs, is on the market. With cheaper than brand name PPIs, it is unclear whether generic omeprazole is as effective clinically. This study compares generic omeprazole with half-dose esomeprazole, the strongest brand name PPI. The half-dose esomeprazole is in fact cheaper than generic omeprazole. Healthy volunteers will take each medication in turn for 7 days and their stomach acid will be measured while taking each medication. We hypothesize that half-dose esomeprazole is better at suppressing stomach acid than generic omeprazole.

ELIGIBILITY:
Inclusion Criteria:

* healthy, non-smoking volunteers older than 18 years of age

Exclusion Criteria:

* history of gastrointestinal disease
* known infection
* previous eradication of Helicobacter pylori
* any prescription or over the counter antacid medication
* pregnant and lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-09; Primary Completion 2017-04 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Median intragastric pH and percentage of time that intragastric pH is above 4 | 24 hours

SECONDARY OUTCOMES:
Nocturnal acid breakthrough, defined as at least 60 continuous minutes of intragastric pH below 4 occurring between 10pm and 6 am and adverse events | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: William G Paterson, MD, Principal Investigator — Queen's University, Hotel Dieu Hospital; Adriana Lazarescu, MD, Principal Investigator — Hotel Dieu Hospital
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada